CLINICAL TRIAL: NCT06684002
Title: Investigation of the Effect of Pilates Exercises on Laxity in Pregnant Women
Brief Title: Effects of Pilates Exercises on Laxity in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcan Suicmez (Other)
Collaborators: Gazi University (Other)
Responsible Party: Sponsor-Investigator, Selcan Suicmez, Sub-Investigator, Ankara Medipol University
Organization: Ankara Medipol University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AnkaraMedipolU-FTR-2024-128
Record Dates: First submitted 2024-11-09; First posted 2024-11-12 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy; Pilates Exercise; Laxity of Ligament
Keywords: pregnancy; laxity; pilates training
MeSH Terms: conditions — Joint Instability | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pilates Group (Experimental): Participants in the Pilates group attended supervised 60-minute sessions twice weekly for eight weeks, led by a certified physiotherapist trained by the Australian Institute of Pilates and Physiotherapy.
  Interventions: Other: Pilates training; Other: Standard prenatal care and ergonomic advice
- Control Group (Other): The control group received standard prenatal care and ergonomic advice, and did not participate in any exercise training.
  Interventions: Other: Standard prenatal care and ergonomic advice

INTERVENTIONS:
Other: Pilates training — Participants in the Pilates group attended supervised 60-minute sessions twice weekly for eight weeks, led by a certified physiotherapist trained by the Australian Institute of Pilates and Physiotherapy.
  Arms: Pilates Group
Other: Standard prenatal care and ergonomic advice — The control group received standard prenatal care and ergonomic advice, and did not participate in any exercise training.

SUMMARY:
The goal of this clinical trial is to investigate whether Pilates exercises can help manage musculoskeletal laxity in pregnant women. It will also examine the safety of Pilates exercises during pregnancy. The primary questions this trial aims to answer are:

Does Pilates exercise reduce the level of laxity in pregnant women? What physical issues do participants experience while performing Pilates exercises during pregnancy?

Participants will:

Engage in Pilates exercises tailored for pregnancy, under the supervision of trained physiotherapists, for a period of 8 weeks.

Attend monthly checkups to monitor progress and record physical health changes. The intention is to determine whether Pilates exercises are effective in improving joint stability and reducing the laxity caused by hormonal changes during pregnancy.

DETAILED DESCRIPTION:
Pregnancy is a physiological process that lasts approximately 40 weeks, during which the embryo completes its development, from fertilization to birth. During this process, significant changes occur in the mother's anatomy, physiology, psychology, and social aspects to maintain maternal homeostasis and ensure optimal fetal growth. The changes during pregnancy are due to four main factors: hormonal-induced changes in collagen tissue and smooth muscle, increased blood volume to enhance circulation to the uterus and kidneys, expansion and displacement of the uterus due to fetal growth, and, lastly, changes in the center of gravity and posture due to weight gain and adaptations. As a result of these changes, pregnant women may experience increases in body weight, ligament laxity, and lumbar lordosis, as well as a decrease in neuromuscular control and abdominal muscle strength, changes in body biomechanics, and a forward shift in the center of gravity. These changes significantly affect the musculoskeletal system, particularly women's bodies. If the body does not adapt to these changes appropriately, potential health problems that threaten the mother's and fetus's health may arise.

Studies have shown that hormonal changes play a role in musculoskeletal system changes from the very beginning of pregnancy. Estrogen, progesterone, endogenous cortisol, and relaxin hormones play significant roles in these changes. Relaxin levels increase until the 12th week of pregnancy, decrease until the 17th week, and stabilize. The increase in relaxin causes tissue relaxation, leading to increased mobility and instability of the pelvic complex and peripheral joints. Estrogen increases in the third trimester and alters bone, cartilage, and ligament structure. Progesterone peaks in the 15th week and induces relaxation effects on muscle structures. These hormonal changes cause physiological relaxation of the pelvic ligaments to facilitate the passage of the fetus through the birth canal. Due to increased levels of relaxin and progesterone, weakened abdominal muscles and an expanding abdomen result in muscle stretching. All of these lead to postural changes, dysfunction in the lumbar and pelvic regions, and weakness in the abdominal muscles. Studies have highlighted that musculoskeletal disorders and increased pain in various joints, such as the knee, observed during pregnancy may be related to laxity.

Regular physical activity has significant benefits for pregnancies that are not complicated by medical or obstetric issues and are classified as low-risk. Therefore, increasing the level of physical activity during pregnancy and performing regular exercises are recommended by the American College of Obstetricians and Gynecologists in their guidelines for physical activity and exercise during pregnancy and the postpartum period. The benefits of regular physical activity and exercise during pregnancy include maintaining and improving physical fitness, preventing excessive gestational weight gain, reducing the risk of pre-eclampsia and preterm birth, decreasing the prevalence of back pain, improving sleep quality, reducing anxiety and depressive symptoms, and enhancing health perception and body image. Due to these beneficial effects, engaging in at least 30 minutes of moderate aerobic exercise five days a week is recommended. However, it has been reported that approximately 15% of women during pregnancy meet the minimum physical activity recommendation (at least 150 minutes of moderate physical activity per week).

Pilates is an exercise method developed by Joseph Hubertus Pilates that activates all the muscular functions of the body, increasing the endurance, flexibility, and strength of all body muscles, particularly the core, and improving balance systems. It also enhances dynamic postural control. The core is the center of the kinetic chain and is responsible for power transfer between the upper and lower body. All movements begin with the contraction of the muscles in the core, and the power generated by these contractions is transferred to the limbs. The core muscles are described as an anatomical box comprising several muscle groups. Over time, the demand for physical therapy to develop the core has increased. Pilates and core exercises, which have proven effectiveness, are among the interventions used for this purpose.

Joseph Pilates, who developed over 600 exercises suitable for various levels and body types, aimed to improve the stabilization of the core muscles-multifidus, transversus abdominis, pelvic floor, and diaphragm muscles, which represent the powerhouse in Pilates-and to improve the strength, endurance, and flexibility of the muscles, ligaments, and fascia that transmit the power generated by these muscles throughout the body, thus promoting overall body health.

Craig Phillips, a physiotherapist and former ballet dancer, led the establishment of the Australian Physiotherapy and Pilates Institute (APPI) and worked to modify Pilates exercises to be more suitable for body biomechanics. Today, modified Pilates, performed by physiotherapists, has emerged as clinical Pilates. This allows physiotherapists to apply Pilates exercise programs tailored to individuals based on clinical Pilates and scientific foundation principles, including for pregnant women.

Clinical Pilates positively affects both maternal health and the health of the fetus. Clinical Pilates is adequate during pregnancy in controlling breathing, improving spinal stabilization, pelvic floor control, and developing proper posture. It also increases muscle tone and strength. Strengthened and developed muscles improve women's activity levels, coordination, and balance. Those who practice Pilates daily experience increased energy throughout the day. Pilates during pregnancy helps restore the balance sense disturbed by postural and hormonal changes, increases joint range of motion and flexibility, and improves strength. It allows women to adapt more comfortably to the temporary body changes that come with pregnancy and move freely with their bodies. Therefore, clinical Pilates is considered an ideal form of exercise for pregnancy.

Considering the changes occurring during pregnancy and the positive effects of Pilates exercises on body systems during pregnancy, it is thought that the effect of Pilates exercises on laxity in pregnant women should be investigated. Therefore, the aim of our study is to examine the effect of the Pilates exercise method on laxity.

In line with our objectives, our hypotheses are as follows:

H0: Pilates exercises have no effect on laxity in pregnant women. H1: Pilates exercises have an effect on laxity in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-35 years
* In the 14th-16th week of pregnancy
* Voluntary participation in the study

Exclusion Criteria:

* Cardiovascular or pulmonary diseases
* Contraindications to exercise during pregnancy
* Prior participation in structured physical activity programs

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 42 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Ligament laxity | 10 minutes
  The anterior tibial translation of the knee will be considered as representative of the anterior laxity of the knee of women measured with an arthrometer ® (bilateral examination repeated 3 times on each knee).The degree of laxity will be evaluated thanks to the international classification IKDC.

SECONDARY OUTCOMES:
Generalized joint hypermobility | 2 minutes
  Generalized joint hypermobility (GJH) was assessed using the Beighton scoring system, which consists of five bilateral and unilateral maneuvers. Each positive test scored one point, with a maximum score of 9. A score of ≥5 indicated GJH.
Physical activity level | 7 days
  Participants' physical activity was monitored using the Omron HJ-321-E pedometer (Omron Healthcare, Japan), which detects vertical oscillations and stores up to seven days of data.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Medipol University, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bulguroglu M, Bulguroglu HI, Degirmenci B, Suicmez S, Gevrek Aslan C, Zorlu Develik S, Atalay Guzel N. Effectiveness of a prenatal pilates program on ligamentous laxity and joint hypermobility in pregnant women: a dual-center randomized controlled trial. BMC Pregnancy Childbirth. 2025 Aug 28;25(1):897. doi: 10.1186/s12884-025-08082-1. PMID 40877820